CLINICAL TRIAL: NCT03414710
Title: A Randomized Controlled Trial Evaluating Efficacy of Promoting Voluntary Medical Male Circumcision Among Male Sexually Transmitted Diseases Patients in China
Brief Title: A RCT Promoting Voluntary Medical Male Circumcision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Zixin Wang, Research Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 81373054
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Behavior, Health
Keywords: uptake of voluntary medical male circumcision
MeSH Terms: conditions — Health Behavior | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Health education booklet plus video plus brief counseling
  In addition to the educational booklet received by the control group, the intervention group will receive the following health promotion:
  1. Watch a 10-minute video promoting VMMC
  2. Receive a brief counseling promoting VMMC If the participants are willing to take up VMMC, the counselors will facilitate them to make an appointment for check-up and surgery.
  Interventions: Behavioral: Health education booklet plus video plus brief counseling
- Control group (Active Comparator): Health education booklet only After randomization took place, the control group will receive an education booklet introducing voluntary medical male circumcision.
  If the participants are willing to take up VMMC, the counselors will facilitate them to make an appointment for check-up and surgery.
  Interventions: Behavioral: Health education booklet only

INTERVENTIONS:
Behavioral: Health education booklet plus video plus brief counseling — Participants in the intervention group will receive a health education booklet, watch a 10-minute video and receive counseling provided by the clinicians
  Arms: Intervention group
Behavioral: Health education booklet only — Participants in the intervention group will only receive a health education booklet
  Arms: Control group

SUMMARY:
A parallel-group, non-blinded randomized controlled trial was conducted. Participants were uncircumcised heterosexual male sexually transmitted disease patients attending the four collaborative public sexually transmitted diseases clinics in three Chinese cities. Those who were known to be HIV positive were excluded. After completion the baseline face-to-face interview, 238 participants will be randomized 1:1 into the intervention group and the control group. Participants in the control group will receive a health education booklet introducing voluntary medical male circumcision. In addition to the health education booklet received by the control group, the intervention group watched a 10-minute video and received a brief counseling delivered by the clinicians. Participants will be followed up by telephone six months afterwards.

DETAILED DESCRIPTION:
Study Design A parallel-group and non-blinded RCT is conducted. Face-to-face interview is conducted at baseline in the collaborating STD clinics. A 5-minute telephone survey is conducted six months afterwards by blinded interviewers. Up to five calls will be made at different timeslots during weekdays/weekends before considering a case as loss-to-follow up.

Participants Inclusion criteria are: 1) Chinese male aged ≥18 years, 2) uncircumcised, 3) diagnosis of any one of the five types of STDs listed in the national surveillance system: Primary, secondary or latent syphilis (determined by Treponemapallidum Particle Assay and Toluidine Red Untreated Serum Test), genital warts (diagnosed by presence of clinical symptoms and supported by biopsy), genital herpes (diagnosed clinically, supported by ELISA), or gonorrhea or NGU (diagnosed by using Polymerase Chain Reaction), and 4) willingness to leave contact information (mobile and/or electronic) with the investigators and be followed up at Month 6. Men who had ever had oral or anal sex with men and those who were known to be HIV positive are excluded.

Recruitment procedures To avoid selection bias, all male sexually transmitted disease patients (MSTDP) attending the five participating clinics during the study period are invited to participate in the study. A clinician ensures the eligibility of the prospective participants to join the study in a consultation room and refers them to the trained counselors who are STD clinicians. The interviewers then brief the participants about the study, assure them that refusals would not affect their right to use any services and that they can quit any time without being questioned. Written informed consent will be sought. Ethics approval was obtained from the Ethics Committee of Guangdong Provincial Dermatology Hospital, Guangzhou, China.

The baseline survey and random allocation process After completion the baseline face-to-face interview, participants will be randomized 1:1 to either the intervention group or the control group. Computer-generated random allocation codes are produced and sealed in opaque envelopes by a research staff with no involvement in recruitment or baseline survey. One envelope will be drawn and opened in front of the participant by the counselors. The counselors then inform the participant which group he is assigned to. Block randomization with block size of eight is used.

The Control Group After randomization took place, the control group will receive an education booklet introducing voluntary medical male circumcision. The contents include: 1) harms of STD infection on men and their female sex partners (e.g., STD infection increases risk of HIV acquisition), 2) benefit of VMMC in reducing risk of HIV and STD infection in men, and the indirect protective effects for their female sex partners, 3) basic information of VMMC, including cost, hospitals that offer VMMC, common side effects and recovery time. If the participants are willing to take up VMMC, the counselors will facilitate them to make an appointment for check-up and surgery.

The Intervention Group

In addition to the educational booklet received by the control group, the intervention group will receive the following health promotion:

1. Watch a 10-minute video promoting VMMC: in the video, a well-known STD clinician talks about severity of STD infection and benefits of VMMC, and gave reminders about the importance of consistent condom use even after taking up VMMC. He also expresses his support to the participants for taking up VMMC. One MSTDP who had taken up VMMC presented a testimonial in the video about his positive experience with VMMC, including mild pain and surgical complications of VMMC, improvement in sexual pleasure and sexual functioning after taking up VMMC, and support received from his peers and female sex partners with respect to VMMC.
2. Receive a brief counseling promoting VMMC: the counselors would discuss with those who consider taking up VMMC about their concerns, and encourage them to make a specific plan to take up VMMC; the counselors also remind those who show no intention to take up VMMC in the next six months about the risk of HIV/STD infection and the benefit of taking up VMMC. If the participants are willing to take up VMMC, the counselors will facilitate them to make an appointment for check-up and surgery.

Measures Outcomes and confounders Potential confounders include socio-demographics, utilization of HIV/STD prevention services, STD history, foreskin condition and condomless sex with regular female sex partners (RP: defined as their wives or stable girlfriends), female sex workers (FSW: defined as a female who exchanged sex for money) and non-regular female sex partners (NRP: defined as a female who was neither FSW nor RP) since exhibiting STD symptoms or receiving an STD diagnosis. The primary outcome was whether the participant has taken up VMMC within the 6-month follow-up period. Secondary outcomes are perceptions related to VMMC based on the Theory of Planned Behavior (scores of the Positive Attitude Scale, the Negative Attitude Scale, the Subjective Norm Scale and the Perceived Behavioral Control Scale).

Process evaluation Process evaluation of health promotion will also be conducted at Month 6. Participants in both groups will be asked: 1) whether the content of the health promotion is clear, 2) whether the materials (video or booklet) is attractive to them, 3) whether the health promotion has increased their understanding about the benefit of VMMC and willingness to take up VMMC. Participants in the intervention group are asked an additional question about their satisfaction of the counseling session.

Post-surgical experience At Months 6, circumcised participants will be asked whether they have any surgical complication, and whether they have sought medical consultation due to such complications. Sexually active circumcised participants will be asked whether they have reduce condom use with RP, NRP or FSW, or increase number of such female sex partners after taking up VMMC.

Sample size planning In a single-arm, non-blinded test-of-concept trial, 19.9% had taken up VMMC during the 4-month follow-up period after exposing to a similar intervention (i.e., watching a 10-minute video clip and receiving brief consultation and a health education booklet). In this study, assuming 20% of the participants will take up VMMC in the intervention group within the 6-month follow period, the sample size of 71 per group would allow us to detect a between-group difference in the uptake of VMMC of 15% or above (a=0.05, 2-sided test with statistical power of 0.8; PASS). Taking into account an expected drop-out rate of 40% at Month 6, a sample size of 119 per group was required. The total sample size would be 238.

Statistical analysis Baseline between-group differences will be compared by using Chi-square test. Intention-to-treat analysis will be used for outcome analyses. Relative risk (RR), absolute risk reduction (ARR), and number needed to treat (NNT) statistics will be used to test between-group difference in primary outcome. Wilcoxon signed-ranked test will be used to test the between-group difference in secondary outcomes. Within-group difference will be tested by using McNemar test. SPSS version 16.0 will be used, and p values <0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Chinese male aged ≥18 years
* uncircumcised
* diagnosis of any one of the five types of STDs listed in the national surveillance system: Primary, secondary or latent syphilis (determined by Treponemapallidum Particle Assay and Toluidine Red Untreated Serum Test), genital warts (diagnosed by presence of clinical symptoms and supported by biopsy), genital herpes (diagnosed clinically, supported by ELISA), or gonorrhea or NGU (diagnosed by using Polymerase Chain Reaction)
* willingness to leave contact information (mobile and/or electronic) with the investigators and be followed up at Month 6

Exclusion Criteria:

* Men who had ever had oral or anal sex with men
* known to be HIV positive

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 244 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Uptake of voluntary medical male circumcision | 6 months
  At month 6, participants will be asked whether they have taken up voluntary medical male circumcision within the 6-month follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Zixin Wang, PhD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Centre for Health Behaviours Research, the Chinese University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Wang Z, Yang L, Hao C, Jiang H, Zhu J, Luo Z, Zheng Z, Lau JTF. A Randomized Controlled Trial Evaluating Efficacy of a Brief Setting-Based and Theory-Based Intervention Promoting Voluntary Medical Male Circumcision Among Heterosexual Male Sexually Transmitted Disease Patients in China. AIDS Behav. 2019 Sep;23(9):2453-2466. doi: 10.1007/s10461-019-02610-9. PMID 31321636